CLINICAL TRIAL: NCT05220904
Title: A Randomized Controlled Clinical Study of Perceptual Learning Improving Visual Function in Patients With Keratoconus
Brief Title: Perceptual Learning Improve Visual Function in Patients With Keratoconus
Acronym: KPL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021KYPJ203
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2023-11

CONDITIONS: Keratoconus, Stable
MeSH Terms: conditions — Keratoconus | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator:placebo practice+spectacles (Placebo Comparator): Patients will take placebo practices with spectacles every two days.
  Interventions: Device: spectacles
- Experimental： perceptual learning practice+spectacles (Experimental): Patients will take perceptual learning practices with spectacles every two days.
  Interventions: Device: spectacles; Device: perceptual learning

INTERVENTIONS:
Device: spectacles — Spectacle is the the most common treatment for refractive errors.
Device: perceptual learning — Blurred vision from the eyes can be improved by enhancing the brain's visual processing.
  Arms: Experimental： perceptual learning practice+spectacles

SUMMARY:
This project aims at non-progressive keratoconus patients with unsatisfactory visual acuity corrected by spectacles, and explores the effectiveness and maintenance of visual acuity improved by perceptual learning.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 9 years or older;
2. Has been diagnosed as Keratoconus,BAD-D≥2.6;
3. Change of Kmax < 1.0 D and change of BAD-D <0.4175 betweem the last two Pentacam result;
4. The best corrected visual acuity of both eyes was between 0.1 and 1.0;
5. Has voluntarily agreed to participate in the study by signing the statement of informed consent.

Exclusion Criteria:

1. Has history of acute keratoconus;
2. Has other eye diseases or other diseases/conditions causing vision loss;
3. Has eye surgery history in the past 1year;
4. Is currently using local/systemic medications or other interventions that may affect visual function;
5. Receiving other treatments that may affect the results of this study, such as contact lenses during the study;
6. Has any known neurological diseases;
7. Participating in other studies currently that may affect the results of this study;
8. Study other reasons that the physician considers inappropriate for inclusion in the program.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-02-05 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
3-months corrected visual acuity | baseline；3 months.
  Mean changes of best corrected visual acuity between 3 months after perceptual learning training and baseline values.

SECONDARY OUTCOMES:
corrected visual acuity of other time frame | 6,9,15 months
  Mean changes of best corrected visual acuity for 6,9,15 months.
ucorrected visual acuity (UCVA) | 3,6,9,15 months
  Mean changes of ucorrected visual acuity (UCVA) for 3,6,9,15 months.
contrast sensitivity function (CSF) | 3,6,9,15 months
  Mean changes of contrast sensitivity function (CSF) for 3,6,9,15 months.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Yang, Professor, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China